CLINICAL TRIAL: NCT05448105
Title: My Diabetes Care: A Scalability and Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, William Martinez, MD, MS, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 220629; R01DK131129 (NIH)
Record Dates: First submitted 2022-06-23; First posted 2022-07-07 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Self-efficacy; Patient Web Portals
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- My Diabetes Care (MDC) (Experimental): Patients have access to a patient web portal embedded with the My Diabetes Care (MDC) intervention.
  Interventions: Other: My Diabetes Care (MDC)

INTERVENTIONS:
Other: My Diabetes Care (MDC) — My Diabetes Care (MDC) is a multi-faceted patient portal intervention that is designed to help patients better understand their diabetes health data as well as promote and support self-management. MDC uses infographics to facilitate patients' understanding of their diabetes health data (e.g., HbA1c, LDL) and provides literacy level-appropriate diabetes self-care information. In this study, the MDC user-interface was expanded to display additional diabetes health-data, including urine microalbumin and weight/body mass index (BMI) and a Spanish-language version of MDC was available to Spanish-speaking patients with limited English proficiency.
  Other Names: Patient-facing Diabetes Dashboard

SUMMARY:
The purpose of this study is to conduct a prospective, longitudinal study on the My Diabetes Care (MDC) mobile intervention to assess usage patterns, user experience, and to uncover errors in functionality prior to a larger interventional trial.

DETAILED DESCRIPTION:
Up to 90 adult patients with type 2 diabetes mellitus will be enrolled and given access to My Diabetes Care (MDC). My Diabetes Care (MDC) is a multi-faceted patient portal intervention for mobile devices that is designed to help patients better understand their diabetes health data as well as promote and support self-management. MDC uses infographics to facilitate patients' understanding of their diabetes health data (e.g., HbA1c, LDL) and provides literacy level-appropriate and tailored diabetes selfcare information. Patients will be invited by mail to be screened for enrollment in the study. Interested patients will be able to complete an electronic consent form and enroll online via Research Electronic Data Capture (REDCap) version 5.0.8. Study participants will complete questionnaires electronically via email using REDCap at two time points: baseline (T0) and one-month follow-up (T1). Participants will complete a baseline questionnaire (T0) including basic demographic questions, items about computer usage and internet access, and validated measures of health literacy and eHealth literacy. Each participant will have access to MDC for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* Age 18-75 years old
* Currently taking at least one medication for diabetes
* Patient at a participating clinic within Vanderbilt Medical Center or Brigham and Women's Hospital
* Able to speak and read in English or Spanish
* Reliable access to a smartphone or tablet with internet access
* Active patient web portal account (for example, My Health at Vanderbilt or Patient Gateway)

Exclusion Criteria:

* Have a medical condition that affects your memory or ability to think
* Have severe difficulty seeing or hearing
* Have a medical condition that makes it hard for people to understand what you are saying

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Martinez, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published in a peer-reviewed journal, de-identified individual participant data that underlie the results reported will be available upon requests made to the principal investigator and ending after 36 months after publication.
Supporting Information: Study Protocol, SAP
Time Frame: Deidentified individual participant data that underlie the results reported will be available after publication in a peer-reviewed journal and posted on clinical trials and ending after 36 months of publication.
Access Criteria: Researchers should provide a methodologically sound proposal to achieve their proposed aims. Proposals may be submitted to the principal investigator up to 36 months following publication. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the enrolled participants, 63 completed the baseline questionnaire and were then assigned to the intervention.
Groups:
- My Diabetes Care (MDC): Patients have access to a patient portal embedded with the My Diabetes Care (MDC) intervention.
  MDC is a multi-faceted patient portal intervention that is designed to help patients better understand their diabetes health data as well as promote and support self-management. MDC uses infographics to facilitate patients' understanding of their diabetes health data (e.g., HbA1c, LDL) and provides literacy level-appropriate diabetes self-care information. In this study, the MDC user-interface was expanded to display additional diabetes health-data, including urine microalbumin and weight/body mass index (BMI) and a Spanish-language version of MDC was available to Spanish-speaking patients with limited English proficiency.
Period: Overall Study
Arm/Group | My Diabetes Care (MDC)
Started | 63
Completed | 63
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- My Diabetes Care (MDC): Patients have access to a patient web portal embedded with the My Diabetes Care (MDC) intervention.
  MDC is a multi-faceted patient portal intervention that is designed to help patients better understand their diabetes health data as well as promote and support self-management. MDC uses infographics to facilitate patients' understanding of their diabetes health data (e.g., HbA1c, LDL) and provides literacy level-appropriate diabetes self-care information. In this study, the MDC user-interface was expanded to display additional diabetes health-data, including urine microalbumin and weight/body mass index (BMI) and a Spanish-language version of MDC was available to Spanish-speaking patients with limited English proficiency.
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (12.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 36
  Male | 26
  Other | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White or Caucasian | 41
  Black or African American | 18
  More than one race | 2
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 63
Language [Count of Participants; unit: Participants]
  English | 57
  Spanish | 6

OUTCOME MEASURES:

1. Primary Outcome: Usability
Description: The System Usability Scale (SUS) is a valid measure of usability and assesses users' perceptions of ease of use, likability of the interface, and overall satisfaction using a 5- point Likert scale (strongly disagree to strongly agree). The ten items are scored on a five-point Likert scale. The item scores are summed and then converted to a score ranging from 0 (worst) to 100 (best). Based on prior research, a score above 68 would be above average and a score of 71 or above suggests 'good' usability.
Time Frame: One month follow-up (t1)
Population: 47 participants used to the study intervention during the study period and completed the SUS scale.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 47
score on a scale | 75.0 [67.5 to 85.0]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Superiority; p = 0.02, Wilcoxon signed rank test; Wilcoxon signed rank test comparing the participants' SUS scores to the threshold value of 71 indicative of "good" usability

2. Primary Outcome: System Usage
Description: System usage will be assessed by user analytics data capturing participant use to MDC during the study period. MDC use is defined as one or more visits to the MDC site during the study period.
Time Frame: One month follow-up (t1)
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 63
Participants
  Yes | 49
  No | 14

3. Primary Outcome: User Experience - Acceptance
Description: User experience will be assessed by study-specific survey items administered to all study participants at the end of the study period (T1). Survey items will assess agreement on a 5-point Likert scale from Strongly Agree to Strongly Disagree. Participants will be asked whether they would continue to use My Diabetes Care (MDC) going forward were it to remain available and whether they would recommend MDC to other patients with diabetes.
Time Frame: One month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period and participants who responded to the items below on the one month follow-up questionnaire (t1).
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
Participants
  Would recommend the intervention to other patients: Strongly agree/ agree | 42
  Would recommend the intervention to other patients: Neutral/ disagree/ strongly disagree | 7
  Would continue to use the intervention in future if it remained available: number analyzed (Participants) | 47
  Would continue to use the intervention in future if it remained available: Strongly agree/ agree | 37
  Would continue to use the intervention in future if it remained available: Neutral/ disagree/ strongly disagree | 10

4. Secondary Outcome: Change in Diabetes Knowledge
Description: The Revised Brief Diabetes Knowledge Test (DKT2) is a valid measure of diabetes knowledge. The 14-item questionnaire was designed to assess a patient's understanding of diabetes management. The DKT2 is a uni-dimensional, 14-item scale with scores ranging from 0 to 14 (number of items answered correctly). Higher scores indicate greater knowledge.
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period and completed the Short Diabetes Knowledge Instrument (SDKI) on the baseline (t0) and one-month follow-up (t1) questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
score on a scale
  baseline questionnaire (t0) | 12.0 [10.0 to 13.0]
  one-month follow-up questionnaire (t1) | 12.0 [11.0 to 14.0]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Other; p = 0.04, paired Wilcoxon signed-rank sum test

5. Secondary Outcome: Change in Diabetes Self-Care - Diet Adherence
Description: The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: diet (4 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The general diet subscale is used to assess diet adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. An example item includes "How many of the last SEVEN DAYS have you followed a healthful eating plan?" The general diet subscale score is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period and completed the Summary of Diabetes Self-Care Activity (SDSCA) scale diet subdomain on the baseline (t0) and one-month follow-up (t1) questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
score on a scale
  baseline (t0) questionnaire | 4.0 [2.8 to 5.0]
  one-month follow-up (T1) questionnaire | 4.8 [3.5 to 5.5]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Other; p < 0.01, paired Wilcoxon signed-rank sum test — This is calculated p-value. The threshold for significance was less than 0.05

6. Secondary Outcome: Change in Diabetes Self-Care - Exercise Adherence
Description: The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: diet (4 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The exercise subscale is used to assess exercise adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. The exercise subscale score is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period and completed the Summary of Diabetes Self-Care Activity (SDSCA) scale exercise subdomain on the baseline (t0) and one-month follow-up (t1) questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
score on a scale
  baseline (t0) questionnaire | 2.0 [0.5 to 3.5]
  one-month follow-up (T1) questionnaire | 2.0 [1.0 to 4.0]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Other; p = 0.16, paired Wilcoxon signed-rank sum test

7. Secondary Outcome: Change in Diabetes Self-Care - Glucose Self-monitoring Adherence
Description: The Summary of Diabetes Self-Care Activity (SDSCA) is a 10-item multidimensional instrument to assess levels of diabetes self-care across five domains: diet (4 items), exercise (2 items), foot care (2 items), and blood-glucose testing (2 items). The blood-glucose testing subscale is used to assess glucose self-monitoring adherence. The instrument is based on the self-reported days completing recommended activities during the past 7 days. The blood-glucose testing subscale score is the mean number of days for the 2 items in the subscale. The score range is from 0 days (worst) to 7 days (best).
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
score on a scale
  baseline (t0) questionnaire | 4.0 [2.5 to 6.0]
  one-month follow-up (T1) questionnaire | 4.0 [2.0 to 6.5]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Other; p = 0.69, paired Wilcoxon signed-rank sum test

8. Secondary Outcome: Change in Diabetes Self-Efficacy
Description: The Perceived Diabetes Self-Management Scale (PDSMS) is a valid measure of diabetes self-efficacy (i.e., how confident they feel about their ability to carry out multiple self management tasks). The uni-dimensional, 8-item scale is scored on a five-point Likert scale. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes.
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period and completed the Perceived Diabetes Self-Management Scale (PDSMS) on the baseline (t0) and one-month follow-up (t1) questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
score on a scale
  baseline questionnaire (t0) | 25.0 [23.0 to 26.0]
  one-month follow-up questionnaire (t1) | 25.0 [23.0 to 27.0]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Other; p = 0.90, paired Wilcoxon signed-rank sum test

9. Secondary Outcome: Change in Medication Adherence
Description: The Adherence to Refills and Medications Scale is a reliable and valid measure of medication adherence. The 12-item scale has item responses range that from 1="none of the time" to 4="all of the time." Responses are summed to produce an overall adherence score ranging from 12-48, with higher scores representing more problems with medication adherence.
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period and completed the Adherence to Refills and Medications Scale on the baseline (t0) and one-month follow-up (t1) questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
score on a scale
  baseline questionnaire (t0) | 15.0 [12.0 to 18.0]
  one-month follow-up questionnaire (t1) | 15.0 [13.0 to 16.5]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Other; p = 0.11, paired Wilcoxon signed-rank sum test

10. Secondary Outcome: Change in Diabetes Distress
Description: The Problem Areas in Diabetes Scale (PAID-5) is a valid measure of diabetes distress. The five-item, uni-dimensional scale has scores that range from 0 to 20, with higher scores suggesting greater diabetes-related emotional distress. The PAID-5 is associated with measures of depression and hemoglobin A1c.
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period and completed the Problem Areas in Diabetes Scale (PAID-5) on the baseline (t0) and one-month follow-up (t1) questionnaires.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
score on a scale
  baseline questionnaire (t0) | 6.0 [3.0 to 10.0]
  one-month questionnaire follow-up (t1) | 5.0 [2.0 to 8.0]
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Test type: Other; p = 0.22, paired Wilcoxon signed-rank sum test

11. Secondary Outcome: Change in Knowledge of Diabetes Measures
Description: Unique study specific items to assess participants' knowledge of measures of diabetes health status (i.e., hemoglobin A1C, blood pressure, low-density lipoprotein, urine microalbumin, and body mass index). Each item has 1 correct answer and several incorrect answers.
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis was limited to participants that used MDC during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
Participants
  Pre-Intervention (t0): Definition of A1c?: Correct | 47
  Pre-Intervention (t0): Definition of A1c?: Incorrect | 2
  Pre-Intervention (t0): Goal range for A1c?: Correct | 27
  Pre-Intervention (t0): Goal range for A1c?: Incorrect | 22
  Pre-Intervention (t0): Definition of systolic blood pressure?: number analyzed (Participants) | 48
  Pre-Intervention (t0): Definition of systolic blood pressure?: Correct | 24
  Pre-Intervention (t0): Definition of systolic blood pressure?: Incorrect | 24
  Pre-Intervention (t0): Goal range for systolic blood pressure?: Correct | 16
  Pre-Intervention (t0): Goal range for systolic blood pressure?: Incorrect | 33
  Pre-Intervention (t0): Definition of LDL cholesterol?: Correct | 30
  Pre-Intervention (t0): Definition of LDL cholesterol?: Incorrect | 19
  Pre-Intervention (t0): Goal range for LDL cholesterol?: Correct | 18
  Pre-Intervention (t0): Goal range for LDL cholesterol?: Incorrect | 31
  Pre-Intervention (t0): Definition of urine microalbumin?: Correct | 28
  Pre-Intervention (t0): Definition of urine microalbumin?: Incorrect | 21
  Pre-Intervention (t0): Goal range for urine microalbumin?: Correct | 13
  Pre-Intervention (t0): Goal range for urine microalbumin?: Incorrect | 36
  Pre-Intervention (t0): Definition of BMI?: Correct | 46
  Pre-Intervention (t0): Definition of BMI?: Incorrect | 3
  Pre-Intervention (t0): Goal range for BMI?: Correct | 18
  Pre-Intervention (t0): Goal range for BMI?: Incorrect | 31
  Post-Intervention (t1): Definition of A1c?: Correct | 46
  Post-Intervention (t1): Definition of A1c?: Incorrect | 3
  Post-Intervention (t1): Goal range for A1c?: Correct | 30
  Post-Intervention (t1): Goal range for A1c?: Incorrect | 19
  Post-Intervention (t1): Definition of systolic blood pressure?: Correct | 31
  Post-Intervention (t1): Definition of systolic blood pressure?: Incorrect | 18
  Post-Intervention (t1): Goal range for systolic blood pressure?: Correct | 19
  Post-Intervention (t1): Goal range for systolic blood pressure?: Incorrect | 30
  Post-Intervention (t1): Definition of LDL cholesterol?: Correct | 37
  Post-Intervention (t1): Definition of LDL cholesterol?: Incorrect | 12
  Post-Intervention (t1): Goal range for LDL cholesterol?: Correct | 23
  Post-Intervention (t1): Goal range for LDL cholesterol?: Incorrect | 26
  Post-Intervention (t1): Definition of urine microalbumin?: Correct | 33
  Post-Intervention (t1): Definition of urine microalbumin?: Incorrect | 16
  Post-Intervention (t1): Goal range for urine microalbumin?: Correct | 16
  Post-Intervention (t1): Goal range for urine microalbumin?: Incorrect | 33
  Post-Intervention (t1): Definition of BMI?: Correct | 45
  Post-Intervention (t1): Definition of BMI?: Incorrect | 4
  Post-Intervention (t1): Goal range for BMI?: Correct | 23
  Post-Intervention (t1): Goal range for BMI?: Incorrect | 26
Statistical Analysis 1: Comparison: My Diabetes Care (MDC); Analysis for pre-post change in knowledge of definition of A1C; Test type: Other; p = 1.00, McNemar — This is the calculated p-value
Statistical Analysis 2: Comparison: My Diabetes Care (MDC); Analysis for pre-post change in knowledge of goal range for hemoglobin A1c; Test type: Other; p = 0.55, McNemar
Statistical Analysis 3: Comparison: My Diabetes Care (MDC); Analysis for pre-post change in knowledge of definition of systolic blood pressure; Test type: Other; p = 0.11, McNemar
Statistical Analysis 4: Comparison: My Diabetes Care (MDC); Analysis of pre-post change in knowledge of goal range for systolic blood pressure; Test type: Other; p = 0.63, McNemar
Statistical Analysis 5: Comparison: My Diabetes Care (MDC); Analysis of pre-post change in knowledge of definition of LDL cholesterol; Test type: Other; p = 0.12, McNemar
Statistical Analysis 6: Comparison: My Diabetes Care (MDC); Analysis for pre-post change in knowledge of goal range for LDL cholesterol; Test type: Other; p = 0.33, McNemar
Statistical Analysis 7: Comparison: My Diabetes Care (MDC); Analysis of pre-post change in knowledge of definition of urine microalbumin; Test type: Other; p = 0.23, McNemar
Statistical Analysis 8: Comparison: My Diabetes Care (MDC); Analysis for pre-post change in knowledge of goal range for urine microalbumin; Test type: Other; p = 0.58, McNemar
Statistical Analysis 9: Comparison: My Diabetes Care (MDC); Analysis of pre-post change in knowledge of definition of body mass index (BMI); Test type: Other; p = 1.00, McNemar
Statistical Analysis 10: Comparison: My Diabetes Care (MDC); Analysis for pre-post change in knowledge of goal range for body mass index (BMI); Test type: Other; p = 0.27, McNemar

12. Secondary Outcome: Change in Diabetes Readiness for Change
Description: Four-item assess the participants' stage of change based on the Transtheoretical Model (TTM) of behavior change including one item each for: (1) physical activity, (2) medication management, (3) glucose self-monitoring, and (4) diet. There are five response options per item that categorize the participants' current TTM stage of change across a continuum: (a) Precontemplation [worst], (b) Contemplation, (c) Preparation, (d) Action, and (e) Maintenance [best]. For each item, precontemplation is represented by the response "No, and I do not intend to in the next 6 months"; contemplation is represented by the response "No, but I am thinking about starting in the next 6 months"; Preparation is represented by the response "No, but I am planning to start in the next 30 days"; action is represented by the response "Yes, I have been for less than 6 months"; and maintenance is represented by the response "Yes, I have been for 6 months or more."
Time Frame: Baseline (t0) to one month follow-up (t1)
Population: Analysis is limited to participants that (1) used MDC during the study period AND (2) completed the survey items at the corresponding timepoints pre-intervention (t0) and post-intervention (T1).
Measure: Count of Participants; unit: Participants
Arm/Group | My Diabetes Care (MDC)
Number analyzed (Participants) | 49
Participants
  Pre-Intervention (t0): Get least 150 minutes of moderate-intensity physical activity per week.: number analyzed (Participants) | 44
  Pre-Intervention (t0): Get least 150 minutes of moderate-intensity physical activity per week.: Precontemplation | 2
  Pre-Intervention (t0): Get least 150 minutes of moderate-intensity physical activity per week.: Contemplation | 7
  Pre-Intervention (t0): Get least 150 minutes of moderate-intensity physical activity per week.: Preparation | 19
  Pre-Intervention (t0): Get least 150 minutes of moderate-intensity physical activity per week.: Action | 5
  Pre-Intervention (t0): Get least 150 minutes of moderate-intensity physical activity per week.: Maintenance | 11
  Post-Intervention (t1): Get least 150 minutes of moderate-intensity physical activity per week.: number analyzed (Participants) | 44
  Post-Intervention (t1): Get least 150 minutes of moderate-intensity physical activity per week.: Precontemplation | 1
  Post-Intervention (t1): Get least 150 minutes of moderate-intensity physical activity per week.: Contemplation | 6
  Post-Intervention (t1): Get least 150 minutes of moderate-intensity physical activity per week.: Preparation | 19
  Post-Intervention (t1): Get least 150 minutes of moderate-intensity physical activity per week.: Action | 11
  Post-Intervention (t1): Get least 150 minutes of moderate-intensity physical activity per week.: Maintenance | 7
  Pre-Intervention (t0): check your blood sugar levels as often as your doctor recommends: number analyzed (Participants) | 43
  Pre-Intervention (t0): check your blood sugar levels as often as your doctor recommends: Precontemplation | 1
  Pre-Intervention (t0): check your blood sugar levels as often as your doctor recommends: Contemplation | 7
  Pre-Intervention (t0): check your blood sugar levels as often as your doctor recommends: Preparation | 6
  Pre-Intervention (t0): check your blood sugar levels as often as your doctor recommends: Action | 10
  Pre-Intervention (t0): check your blood sugar levels as often as your doctor recommends: Maintenance | 19
  Post-Intervention (t1): check your blood sugar levels as often as your doctor recommends: number analyzed (Participants) | 44
  Post-Intervention (t1): check your blood sugar levels as often as your doctor recommends: Precontemplation | 3
  Post-Intervention (t1): check your blood sugar levels as often as your doctor recommends: Contemplation | 1
  Post-Intervention (t1): check your blood sugar levels as often as your doctor recommends: Preparation | 6
  Post-Intervention (t1): check your blood sugar levels as often as your doctor recommends: Action | 12
  Post-Intervention (t1): check your blood sugar levels as often as your doctor recommends: Maintenance | 22
  Pre-Intervention (t0): follow a healthy diet for people with diabetes: number analyzed (Participants) | 44
  Pre-Intervention (t0): follow a healthy diet for people with diabetes: Precontemplation | 2
  Pre-Intervention (t0): follow a healthy diet for people with diabetes: Contemplation | 5
  Pre-Intervention (t0): follow a healthy diet for people with diabetes: Preparation | 12
  Pre-Intervention (t0): follow a healthy diet for people with diabetes: Action | 9
  Pre-Intervention (t0): follow a healthy diet for people with diabetes: Maintenance | 16
  Post-Intervention (t1): follow a healthy diet for people with diabetes: number analyzed (Participants) | 44
  Post-Intervention (t1): follow a healthy diet for people with diabetes: Precontemplation | 0
  Post-Intervention (t1): follow a healthy diet for people with diabetes: Contemplation | 3
  Post-Intervention (t1): follow a healthy diet for people with diabetes: Preparation | 11
  Post-Intervention (t1): follow a healthy diet for people with diabetes: Action | 9
  Post-Intervention (t1): follow a healthy diet for people with diabetes: Maintenance | 21
  Pre-Intervention (t0): take your medicines every day as prescribed: number analyzed (Participants) | 44
  Pre-Intervention (t0): take your medicines every day as prescribed: Precontemplation | 0
  Pre-Intervention (t0): take your medicines every day as prescribed: Contemplation | 0
  Pre-Intervention (t0): take your medicines every day as prescribed: Preparation | 0
  Pre-Intervention (t0): take your medicines every day as prescribed: Action | 3
  Pre-Intervention (t0): take your medicines every day as prescribed: Maintenance | 41
  Post-Intervention (t1): take your medicines every day as prescribed: number analyzed (Participants) | 44
  Post-Intervention (t1): take your medicines every day as prescribed: Precontemplation | 1
  Post-Intervention (t1): take your medicines every day as prescribed: Contemplation | 0
  Post-Intervention (t1): take your medicines every day as prescribed: Preparation | 2
  Post-Intervention (t1): take your medicines every day as prescribed: Action | 2
  Post-Intervention (t1): take your medicines every day as prescribed: Maintenance | 39

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | My Diabetes Care (MDC)
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63
Other Adverse Events (participants affected / at risk) | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/05/NCT05448105/Prot_SAP_001.pdf
  • Informed Consent Form (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT05448105/ICF_000.pdf